CLINICAL TRIAL: NCT07270185
Title: Measuring Outcomes With Validated Exercise
Acronym: MOVE
Status: Recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: H-46255; 99086845 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Physical Activity
Keywords: Wearable accelerometers; COSMED K5 device; Montoye; ActiGraph; SciKit Digital Health (SKDH)
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physical activity assessment in healthy adults: Healthy adults who can meet the eligibility criteria will comprise the study cohort.

SUMMARY:
Physical activity and its intensity level is a critical determinant of health. Digital Health Technologies, such as wearable accelerometers (wrist-worn watch-like devices), can provide researchers and clinicians with objective measures of activity intensity, duration, and effect on an individual's physiology which can provide important insight into overall health. The purpose of this observational study is to assess how well wrist-worn devices can measure the intensity of movement and exercise. This study is designed to rigorously validate existing activity classification algorithms using synchronized multi-sensor data and indirect calorimetry during structured, semi-structured, and free-living tasks.

DETAILED DESCRIPTION:
The study involves three in person visits and a one week at home period with the first visit being an intake assessment of eligibility to participate in the study. If a participant consents to participate and meets inclusion/exclusion criteria, the participant will be scheduled for the follow on in clinic visits. The second visit is the first of two in-laboratory activity-based visits. Healthy participants will wear: 1) three wrist-worn watch-like devices, the ActiGraph CentrePoint Insight Watch (CPIW), the ActiGraph Long-range Energy Alternatives Planning system (LEAP), and the GENEActiv, to measure movement, 2) a portable indirect calorimeter, the COSMED K5 Wearable Metabolic System, to measure oxygen use, 3) a heart rate monitor, the Polar Beat H10, while performing a pre-determined set of physical activities and activities of daily living, which range in intensity from sedentary to vigorous. The pre-determined activities participants will complete during the first physical activity-based visit include treadmill walking and running, posture transitions (e.g., lying, sitting, standing), ambulatory tasks, and activities of daily living which include sweeping with a broom, vacuuming, washing dishes, writing, and folding laundry. Following the completion of the first physical activity in-clinic visit, participants will complete a one week at home period. During the at home portion of the study, participants will be asked to complete the same daily living tasks previously listed, keep a daily activity diary, and wear one wrist-worn watch-like device, the ActiGraph CPIW, on their non-dominant wrist. Upon completion of the one week at home period, participants will complete their third and final in-clinic visit, where the participants will repeat all of the same activities and monitoring of movement through wearing: 1) three wrist-worn watch-like devices, the ActiGraph CPIW, the ActiGraph LEAP, and the GENEActiv, to measure movement, 2) a portable indirect calorimeter, the COSMED K5 Wearable Metabolic System, to measure oxygen use, 3) a heart rate monitor, the Polar Beat H10, while performing a pre-determined set of physical activities and activities of daily living, which range in intensity from sedentary to vigorous.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to comply with study instructions, study visits, and procedures including wearing a tight-fitting respiratory mask
* Able to ambulate independently, including walking/running on a treadmill without assistance.
* Demonstrates fluency in English
* Montreal Cognitive Assessment (MoCA) score of ≥26
* Score of 100 on the Barthel Index
* Participant has reliable access to internet

Exclusion Criteria:

* Participation in other digital device trials within 1 week or investigational drug trials within 5 half-lives of last dose.
* Allergy to polyurethane resin (strap/wristband component), silicone rubber, nickel and/or steel.
* Has any planned surgical, dental, or medical procedure that would overlap with study participation.
* Participants with cardiac pacemakers, electronic pumps or any other implanted medical devices.
* Has any clinically significant medical disorder, condition, disease or clinically significant finding at intake that precludes participant's participation in study activities including any self-reported diagnosis of cardiovascular disease, metabolic disorder, chronic obstructive pulmonary disease, cerebral vascular accident/stroke, stage 2 hypertension, use of any medication which alters heart rate (HR) response (e.g., Beta blockers and calcium blockers), any history of myocardial infarction high-risk unstable angina, uncontrolled cardiac arrhythmias, active endocarditis, symptomatic severe aortic stenosis, decompensated symptomatic heart failure, acute pulmonary embolus or pulmonary infarction, acute noncardiac disorder that my affect exercise performance/be worsened by exercise (e.g., infection, renal failure), acute myocarditis or pericarditis, left main coronary stenosis or its equivalent, moderate stenotic valvular heart disease, electrolyte abnormalities, tachyarrhythmia or bradyarrhythmia's, atrial fibrillation, high-degree Atrioventricular (AV) block, mobility/orthopedic limitations.
* Has any skin conditions, open wounds, or other conditions on the wrists that may interfere with wrist-worn wearable sensors.
* Has tuberculosis, oral lesions (sores, bleeding gums), any respiratory illnesses, and/or any other known transmissible infectious diseases during subsequent study visits.
* Any changes to recorded health status from intake that would deem participant to be ineligible during subsequent study visits.
* Has Asthma
* Has claustrophobia
* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are employees directly involved in the conduct of the study.
* Has a history of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) wine, 12 ounces (360 mL) of beer, or 1.5 ounces (45 mL) of hard liquor) within 12 months of Visit 1 as disclosed by participant during evaluation.
* Is a female who is breastfeeding or pregnant, as disclosed by the participant.
* Class III Obesity: Body Mass Index (BMI) ≥ 40 kg/m2
* Underweight: BMI < 18.5 kg/m2
* Resting systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg
* Resting heart rate <40 or ≥ 110 beats/min (for participants ≥60 years)
* Current tobacco/nicotine use

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will come from patients who receive care at Boston Medical Center or on the Boston University Medical Campus and who reply to posted flyers about the research study. It is anticipated that about 80 healthy interested individuals 18-89 years old (half 18-59 and half 60-89) will be enrolled and after attrition ultimately data from 54 will be analyzed for the sample.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Physical activity (PA) based on algorithms compared to indirect calorimetry | 5 days
  The performance of current physical activity algorithms (e.g. Staudenmayer, SKDH, Montoye) will be compared to indirect calorimetry applied on multiple test devices to estimate physical activity levels.

SECONDARY OUTCOMES:
Consistency of endpoints to assess physical activity | 5 days
  The consistency of endpoints derived by current PA algorithm (e.g. Staudenmayer, SKDH, Montoye) will be compared to one another on multiple wearable Digital health technologies (DHTs) devices.
Reliability of PA algorithms | 5 days
  Test-retest reliability of PA algorithms applied on multiple test devices will be compared with indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD MBA, Principal Investigator — CABUSM, Anatomy and Neurobiology
Locations (1):
- Boston Medical Center and BU Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided